CLINICAL TRIAL: NCT03460873
Title: Prognostic Factor in the Patients With Benign Prostatic Hyperplasia Who Undergo Holmium Laser Enucleation of the Prostate
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, Professor, Samsung Medical Center
Other Study IDs: 2015-11-037
Record Dates: First submitted 2018-02-27; First posted 2018-03-09 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: holmium laser enucleation of the prostate — undergo holmium laser enucleation of the prostate

SUMMARY:
Prognostic factor in the patients with benign prostatic hyperplasia (BPH) who undergo holmium laser enucleation of the prostate

ELIGIBILITY:
Inclusion Criteria:

* Male patient scheduled to undergo prostatectomy using holmium laser

Exclusion Criteria:

* Urethral stricture, large bladder diverticulum, bladder neck contracture

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male patient scheduled to undergo prostatectomy using holmium laser
Study Population: tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Comparison of IPSS(International Prostate Symptom Score) changes | pre-operation and post-operation (3month, 6month)
  Complete the questionnaire(IPSS) before and after the treatment

SECONDARY OUTCOMES:
changes of voided urine volume | pre-operation and post-operation (3month, 6month)
  Comparison of voided urine volume
changes of residual urine volume | pre-operation and post-operation (3month, 6month)
  Comparison of residual urine volume
Occurrence of adverse event | post-operation (3month, 6month)
  collection of adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea